CLINICAL TRIAL: NCT04174820
Title: Child's Study of the Distant Impact of Posterior Fossa Injury on Motor Skills, Language, Cognitive Functioning, and Social Cognition - a Combination of Clinical Assessments and Brain Imaging
Brief Title: Child's Study of the Impact of PF Lesion on Motor Skills, Language, Cognitive Functioning and Social Cognition
Acronym: CervIRM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other); National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 49RC18_0010
Record Dates: First submitted 2019-11-08; First posted 2019-11-22 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Medulloblastoma, Childhood; Healthy Volunteers; Fossa Posterior Tumor; Low-grade Glioma
Keywords: Functional Magnetic Resonance Imaging
MeSH Terms: conditions — Medulloblastoma; Infratentorial Neoplasms | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Retrospective Low-Grade Glioma: Inclusion of patients with Low-Grade Glioma treated one year ago, with functional Magnetic Resonance Imaging, speech therapy, neuropsychological, balance and dexterity tests
  Interventions: Other: Functional Magnetic Resonance Imaging (fMRI)
- Retrospective Medulloblastoma: Inclusion of patients with Medulloblastoma treated one year ago, with functional Magnetic Resonance Imaging, speech therapy, neuropsychological, balance and dexterity tests
  Interventions: Other: Functional Magnetic Resonance Imaging (fMRI)
- Prospective patients: Inclusion of prospective patients with an indication to surgery of a Posterior Fossa Tumor, with evaluation of post-operative mutism and then one year after the end of mutism, an evaluation with functional Magnetic Resonance Imaging, speech therapy, neuropsychological, balance and dexterity tests
  Interventions: Other: Functional Magnetic Resonance Imaging (fMRI)
- Control patients: Inclusion of patients without Posterior Fossa Tumor, with functional Magnetic Resonance Imaging, speech therapy, neuropsychological, balance and dexterity tests
  Interventions: Other: Functional Magnetic Resonance Imaging (fMRI)

INTERVENTIONS:
Other: Functional Magnetic Resonance Imaging (fMRI) — list of the tests: Box and Blocks test, Nine Hole Peg test, walkway GAITRite, EXALang tests, NEPSY II subtests, BRIEF, FEE, WISC 5 tests
  Other Names: Speech Therapy Tests; Neuropsychological Tests; Balance and Dexterity Tests

SUMMARY:
One of the major complications of posterior fossa surgery is Posterior Fossa Syndrome (PFS). This syndrome is due to a possible complication of surgical excision of a tumor of the cerebellum (4th ventricle) and is characterized by transient postoperative mutism, dysarthria, behavioral, and affective disorders, as well as motor disorders. PFS is thought to be related to axonal lesions. The long-term consequences on the cognitive and psychosocial sphere of PFS have been widely documented. On the other hand, the literature concerning the consequences of this syndrome on language is much restricted. Beyond the language, the role of cerebellum would be central in cognition, some authors even comparing it to a great "conductor" who would underlie the learning of most motor and cognitive automatisms.

DETAILED DESCRIPTION:
The physiopathology and the anatomo-functional correlates of motor, cognitive, and language functions after surgery of PF tumors are still rare and little known. The objective of this study is to analyze them via morphometric MRI analysis and functional and structural connectivity in children away from PF surgery, coupled with clinical data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a low grade glioma of the posterior fossa or a medulloblastoma
* Healthy volunteers without any tumor in the posterior fossa (control case)
* At one year of the last treatment for the retrospective groups, or patient who have an indication to a surgery of a tumor of the posterior fossa
* Eligibility to a functional MRI
* Informed consent dated and signed by the holder of the parental authority (if minor) or by the patient (if major) to take part in the study
* Affiliated to a Social Security scheme

Exclusion Criteria:

* Antecedent of neurologic, metabolic or genetic disease
* Brainstem glioma
* Have a contraindication to a MRI

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Case-control study with prospective and retrospective, multicentric recruitment where patients will be included with a low grade glioma of the posterior fossa or a medulloblastoma compared to a healthy volunteers group.
Sampling Method: Non-Probability Sample
Enrollment: 145 (Estimated)
Dates: Start 2020-11-12 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Structural and functional connectives in brain MRI | One day
  Review and compare, in MRI, the structural and functional cerebellar-hemispheric connectives. The primary endpoint the analysis of fMRI brain mapping in accordance to the relations with the motor functions (balance and dexterity), cognitive, behavioral/social cognition and language after treatment for a child's posterior fossa tumor (with or without posterior fossa syndrome) and, in comparison with matched control group on age, sex and level study. The MRI data will be the subject of a specific statistical treatment, via dedicated software, which will be implemented under the control of the investigators who have conducted such an fMRI analysis in previous studies. Various brain mapping can be established from the data collected. It may include statistical comparisons between different preselected regions, and different experimental conditions, or correlation studies between brain activation and clinical parameters.

SECONDARY OUTCOMES:
Dexterity with Box and Blocks test | One day
  Evaluation of the dexterity with Box and Blocks test (number of displaced blocks with each hand).
Dexterity with Nine Hole Peg test | One day
  Evaluation of the dexterity with Nine Hole Peg test (sum of time of realization of the test in seconds and number of displaced pegs).
The balance and the walk | One day
  Evaluation of the balance and the walk with the walkway (time in seconds for the completion of the walkway).
Language functions | One day
  Evaluation of the language functions with the EXALang tests (lexicology, phonology, oral expression, oral understand, reading ...).
Social cognition functions and the cognitive function: recognition of the affects | One day
  Evaluation with the NEPSY II subtests (total score of 35).
Social cognition functions and the cognitive function: behavioural executive functions | One day
  Evaluation with the BRIEF test (86 items for parents).
Social cognition functions and the cognitive function: flexibility | One day
  Evaluation with the FEE test (completion time and number of errors).
Social cognition functions and the cognitive function: perceptual and verbal reasoning | One day
  Evaluation with the WISC V test (number of correct answers).
Patients characteristics | One day
  Age, sociodemographics, personal and cancer history.
Quality of life of patients: PedsQL questionnaire | One day
  Comparison of score of Quality of Life questionnaire (PedsQL 4.0: Pediatric Quality of Life Inventory Version 4.0 Generic Core Scales) between the four groups of the study. The Quality of Life questionnaire PedsQL 4.0 is composed of 23 items comprising 4 dimensions. Items are reversed scored and linearly transformed to a 0-100 scale. In order to get a total score we must sum all the items scores over the number of items answered on all the scales. If more than 50% of the items in the scale are missing, the scale scores should not be computed.

CONTACTS AND LOCATIONS:
Overall Officials: Mickaël Dinomais, MD, Principal Investigator — University Hospital, Angers
Locations (5):
- France (5):
  - CHU Angers, Angers
  - Hôpital Necker, Paris
  - Institut Curie, Paris
  - Hôpitaux Saint-Maurice, Saint-Maurice
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No